CLINICAL TRIAL: NCT07336615
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Impact of CLB101TM️ on Gut Health in Healthy, Overweight Individuals
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: ClostraBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PS22
Record Dates: First submitted 2025-11-18; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal; Overweight , Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Study team
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study product CLB101 (Experimental): Study group will receive the study product CLB101
  Interventions: Dietary Supplement: CLB101™️
- Placebo control (Placebo Comparator): Placebo control group will only receive the placebo until the end of study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: CLB101™️ — CLB101™️ is a probiotic isolated from healthy humans.
  Arms: Study product CLB101
Other: Placebo — Placebo control.
  Arms: Placebo control

SUMMARY:
Anaerostipes caccae CLB101TM️ is a next-generation probiotic isolated from healthy humans. It was shown to be in decreased abundance in people with protein-based food sensitivities/allergies. CLB101TM️ is different from most commercially available probiotics in that it directly produces butyrate. Butyrate is a naturally occurring small molecule found in the gut of healthy individuals, and it has been shown to provide clinical benefits including strengthening the gut lining, providing immune health, and supporting a balanced microbiome. The rationale for developing CLB101TM️ is to provide a probiotic that generates butyrate in the targeted intestinal locations where it can optimally benefit cells that line the gut.

DETAILED DESCRIPTION:
The rationale for this study is to observe the impact of a probiotic supplement called CLB101TM️ on gut health in overweight individuals with moderate to severe gastrointestinal discomfort. Additionally, the study aims to observe the impact of the probiotic product on gastrointestinal symptoms, blood parameters, gut microbiota, as well as its impact on intestinal permeability via activities and technologies that can successfully and effectively be completed and utilized in a home setting. A consumer-driven, decentralized observational clinical research study is therefore well-suited for examining the effects of this probiotic product in this population. The study team will examine the outcomes in a broad age-range of adults who have chosen to try this product. The study will incorporate participant reported outcome questionnaires and surveys and at-home stool collection. There is no "doctor-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the product and take part in the observational process with self-reported measures and at-home sample collection. Findings from this study will contribute knowledge toward the tolerability and formulation of the probiotic product and the design of future studies.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years old, inclusive
* Has self-reported moderate to severe gastrointestinal or digestive symptoms, such as abdominal pain, bloating, flatulence, constipation, or diarrhea.
* Has a Gastrointestinal Symptom Rating Scale (GSRS) score between 4-7.
* Has a Body Mass Index (BMI) >27 but <35.0 kg/m^2.
* Willingness to refrain from taking probiotics or prebiotics during the study period.
* Interested in understanding more about their gut health and the use of probiotic products.
* If taking any OTC or prescription medications for anxiety (e.g. magnesium, anticholinergics, Buspirone, Tricyclics, MAOIs,) or other class of medication for anxiety, must be on a stable dose for at least 4 weeks prior to randomization and throughout the course of the study.
* If using any cannabis-containing products, must be on a stable dose regimen for at least 4 weeks prior to randomization and throughout the course of the study.
* If using any nicotine-containing products, must be on a stable regimen for at least 4 weeks prior to randomization and throughout the course of the study.

Willing to practice a reliable method of contraception for the duration of the study

* In good general health at the time of screening (Investigator discretion).
* Able to read and understand English.
* Able to read, understand, and provide informed consent.
* Able to use a personal smartphone device and download Chloe by People Science.
* Able to receive shipment of the product at an address within the United States and use at-home refrigerator and/or freezer.
* Able to complete study assessments including two stool sample collections, two blood sample collections, two intestinal permeability urine tests, and a food diary over the course of up to 12 weeks.

Exclusion Criteria:

* Participants that do not have a personal smartphone, internet access, or unwilling to download Chloe.
* Participants who are currently on a carnivore diet, raw food diet, fruitarian, liquid diet (does not include vegans or vegetarians).
* Participants receiving any investigational therapies or treatments within 30 days prior to randomization.
* Participants currently taking or have taken antibiotics, probiotic, or prebiotic supplements within the past 4 weeks prior to randomization.
* Participants using immunosuppressive medications, systemic steroids, antifungals, NSAIDs or other medications known to significantly impact gastrointestinal function or microbiota.
* Participants with a clinical diagnosis of any gastrointestinal illness, including but not limited to:
* Inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* Gastroesophageal reflux disease (GERD)
* Gastric or duodenal ulcers
* Celiac disease
* Diverticular disease
* Chronic pancreatitis
* Gastroparesis
* Severe liver disease (e.g., cirrhosis, hepatitis, NAFLD acceptable)
* Gallbladder disease (e.g., cholecystitis, cholelithiasis)
* Gastrointestinal cancer (Colorectal, Intestinal, Stomach, Liver, Gallbladder)
* Participants with a known or suspected gastrointestinal infection, such as:
* Clostridium difficile infection
* Helicobacter pylori infection
* Parasitic infections (e.g., Giardia, Cryptosporidium)
* Participants with a history of gastrointestinal surgery, excluding appendectomy and cholecystectomy.
* Participants with a history of gastrointestinal bleeding or perforation.
* Currently diagnosed with Alcohol Use Disorder and/or Substance Use Disorder.
* Currently pregnant, planning to become pregnant in the next 3 months, or breastfeeding
* Any underlying medical conditions or comorbidities that may confound the assessment of digestive symptoms or the evaluation of the study outcomes.
* Have a significant illness, disease or condition which, in the opinion of the principal investigator, may impact their ability to participate in the study or impact the study outcomes.
* Known hypersensitivity or previous allergic reaction to probiotics, microcrystalline cellulose, vegetarian capsules, silica, or magnesium stearate.
* Are unlikely for any reason to be able to comply with the trial or considered unsuited for participation in the study by the Principal Investigator.
* Consume more than 2 (two) alcoholic drinks per day.
* Cannabis or nicotine use that is weekly or more frequent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and Female
Enrollment: 48 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-03-26 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 6 weeks
  The primary outcome measure is to observe the safety and tolerability of the study product. Assessment of the number, frequency, and severity of adverse events (AEs), serious adverse events (SAEs) and AE withdrawals reported over the study product/placebo use period.

SECONDARY OUTCOMES:
Gastrointestinal Symptoms | 6 Weeks
  A secondary outcome measure will be to assess the impact of the study product. on gastrointestinal symotoms. This will be measured by assessing the change from in Gastrointestinal Symptom Questionnaire score between study product and placebo. The instruments uses a likert scale:
  Absent - I did not have this symptom at all Mild - I had this symptom occasionally, but it did not really bother me Moderate - I had this symptom often, it bothered me quite a bit Severe - I had this symptom very often, it bothered me a great deal), with a lower value indicating a better outcome
Gastrointestinal Symptoms | 6 Weeks
  A secondary outcome measure is to assess the impact of the study product on gastrointestinal symptoms by assessing the change in average scores of gastrointestinal symptoms (i.e., flatulence, bloating, abdominal discomfort, stool consistency/ regularity with modified scale assessment, constipation) between placebo and study product group as measured by a 10-point VAS with 0 being absent and 10 being severe
Blood biomarkers | 6 weeks
  Another secondary outcome is to evaluate the change from baseline in blood blood biomarkers including serum LPS- BP, fecal Calprotectin, Zonulin, Lactoferrin, Butyrate, and ALT/AST at the end of Week 4 between placebo and study product groups.
Gut microbiome | 6 Weeks
  This will be evaluated by looking at the changes from baseline in gut microbiome composition and quantity of A. caccae at Week 4 as analyzed by sequencing and qPRC of stool specimens between study product and placebo groups
Intestinal permeability. | 6 weeks
  Another secondary outcome measure is to evaluate the change from baseline in intestinal permeability at Week 4 as measured by Intestinal Permeability assessment/Leaky Gut Test between placebo and study product groups.

CONTACTS AND LOCATIONS:
Overall Officials: Naoh Craft, MD, Principal Investigator — People Science
Locations (1):
- People Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
This will need to be discussed internally.